CLINICAL TRIAL: NCT07029217
Title: A Prospective Phase III Study Comparing Standard Radiotherapy (24 Gy) With a PET REsponse-guided Very Low Dose (4 Gy) Staged Radiotherapy Strategy for Potentially Curable, Indolent B-cell Lymphomas
Brief Title: A Study of Reduced Dose Radiation Therapy for People With B-Cell Lymphomas
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-089
Record Dates: First submitted 2025-06-10; First posted 2025-06-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma
Keywords: Stage I-II; Radiotherapy; 25-089
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: This a phase III, randomized, multi-center non-inferiority trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Very low dose of Radiation (Active Comparator): Patients will receive a total of 4 Gy in 1-2 consecutive daily fractions comprehensively to all initially involved sites of disease. At 12 weeks (+/- 4 weeks) post VLDRT, the patient will undergo repeat imaging and clinical evaluation.
  Interventions: Radiation: Radiation (Very low dose)
- Standard dose of Radiation (Experimental): Patients will receive a total of 24 Gy in 12 fractions comprehensively to all initially involved sites of disease over 12 consecutive business days. At 12 weeks (+/- 4 weeks) post VLDRT, the patient will undergo repeat imaging and clinical evaluation.
  Interventions: Radiation: Radiation (Standard)

INTERVENTIONS:
Radiation: Radiation (Standard) — 24 Gy in 12 fractions
  Arms: Standard dose of Radiation
Radiation: Radiation (Very low dose) — 4 Gy in 1-2 consecutive daily fractions
  Arms: Very low dose of Radiation

SUMMARY:
The researchers are doing this study to find out whether a very low dose of radiation therapy (VLDRT) is an effective treatment for people with follicular lymphoma (FL) or marginal zone lymphoma (MZL) and works as well as the standard dose of radiation therapy. The researchers will see if VLDRT works against cancer in the area that is currently affected by cancer and if the therapy prevents new spots of lymphoma from developing. The researchers will also compare VLDRT with the standard dose of radiation therapy to see if VLDRT causes fewer side effects.

Radiation therapy uses beams of intense energy to kill cancer cells. Standard doses of radiation therapy can cause short- and long-term side effects. Researchers think VLDRT may be as effective as standard doses, and, because VLDRT uses less radiation, researchers think VLDRT may cause fewer side effects than standard doses.

ELIGIBILITY:
Inclusion Criteria: (Arms 1&2)

* Patients must be diagnosed with a follicular lymphoma or marginal zone lymphoma. Of note, there are now two widely-utilized pathology classification criteria used for mature B-cell lymphomas, the World Health Organization (WHO) 5th Edition Classification of Lymphoid Neoplasms and the International Consensus Classification (ICC) of Mature Lymphoid Neoplasms. Either criteria is acceptable and for the purposes of this protocol, the following diagnoses are included:

  * Follicular lymphoma

    * WHO 5th Edition

      * Classic follicular lymphoma (cFL)
      * Follicular lymphoma with uncommon features (uFL)
      * Pediatric type follicular lymphoma
      * Duodenal type follicular lymphoma
    * ICC

      * Follicular lymphoma, grades 1-2 or 3A
      * BCL2 rearrangement negative, CD23 positive follicle center lymphoma
      * Pediatric type follicular lymphoma
      * Duodenal type follicular lymphoma
  * Marginal zone lymphoma

    * WHO 5th Edition and ICC

      * Nodal marginal zone lymphoma
      * Pediatric nodal marginal zone lymphoma
      * Extranodal marginal zone lymphoma of mucosa associated lymphoid tissue (MALT)
* Patients must have stage I or II disease (with stage I defined as involvement of one nodal region and stage II as two or more nodal regions involved on the same side of the diaphragm)
* Patients should be newly diagnosed or previously observed with no prior lymphoma-directed therapy
* If the patient is referred for localized gastric MALT lymphoma, there should be documented negative H. Pylori testing within 6 months prior to proposed radiotherapy
* Age at the time of enrollment of ≥18 years
* Patients must be able to start radiation within 2 months from time of randomization

Exclusion Criteria:

* Prior radiation to site(s) needing treatment
* Follicular lymphoma, grade 3B (ICC) or Follicular large B cell lymphoma (FLBL by WHO 5th edition criteria)
* Patients planned to receive concurrent systemic therapy (including oral steroids) for their lymphoma
* Patient has cutaneous only iNHL defined as primary cutaneous B-cell lymphoma, primary cutaneous follicle center lymphoma, cutaneous marginal zone lymphoma or unspecified indolent lymphoma of the skin
* Gross total resection of all disease
* Tumor size measuring ≥5 cm in maximum diameter on any modality diagnostic imaging
* Patients with any concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years
  Progression will be defined as either PD as per Lugano criteria (either treated or non-treated lesions) OR
  * Receipt of any additional radiotherapy for lymphoma to an initially involved site outside of the protocol mandated treatment OR
  * Death from any cause

SECONDARY OUTCOMES:
radiographic response | 6 months
  using Lugano criteria

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Imber, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org